CLINICAL TRIAL: NCT00732472
Title: A Randomised, Double-blind, Placebo-controlled, Dose Ascending, 2-cohort, Parallel Group Study to Examine the Safety, Tolerability and Pharmacokinetics of Once-daily Inhaled Doses of GSK573719 Formulated With the Excipient Magnesium Stearatein COPD Subjects for 7 Days
Brief Title: A Study to Assess the Safety and Tolerability of Once Daily Inhaled Doses of GSK573719 Made With Magnesium Stearate in Subjects With Chronic Obstructive Pulmonary Disease(COPD)for 7 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105211
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Magnesium stearate; GSK573719
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 7 day repeat dose (Experimental): 7 day repeat dose
  Interventions: Drug: GSK573719

INTERVENTIONS:
Drug: GSK573719 — 7 day repeat dose

SUMMARY:
The study drug which is an inhaled bronchodilator (lung airway relaxant)has been given to both healthy volunteers and to COPD patients before. This study will assess a new formulation of GSK573719. Many drugs are known to deteriorate over time. To make the study medicine less likely to deteriorate in its container, it is mixed with an inactive substance that helps to to maintain the quality of the study medicine. Previous studies have looked at GSK573719 with another inactive substance called Cellobiose Octaacetate (COA). This study will be looking at a new formulation of GSK573719 using Magnesium Stearate (MgSt) as the inactive substance. MgSt itself is not a medicine but is approved as a food ingredient and has also has been approved to be used in a number of marketed medical inhalers. The purpose of this study is to assess the safety and tolerability of compound GSK573719 with Magnesium Stearate for once-daily treatment of COPD(Chronic Obstructive Pulmonary Disease). This drug will be given to 2 groups of 12 people for 7 days. Group 1 will receive 250mcg or placebo and group 2 will receive 1000mcg or placebo. Group 2 will not be dosed until at least 6 people have completed dosing in group 1 without any significant safety concerns. The following safety measures will be assessed including: ECGs, heart rate, blood pressure, blood samples for safety labs, lung function and 24 hour monitoring of the heart. We will also take blood and urine samples to measure medication levels in the body.

GlaxoSmithKline will be funding the research and it will be recruiting at Synexus in 7 of their centres in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 75 years of age
* A female subject is eligible to participate if she is of:

  * Non childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy, bilateral salpingectomy or bilateral oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Male subjects must agree to use one of the listed contraception methods. This criterion must be followed from the time of the first dose of study medication until 90 days post-last dose.
* Subject diagnosed with COPD, as defined by the GOLD guidelines.
* BMI within the range 18 - 34 kg/m2 (inclusive).
* Subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (Pack years = (cigarettes per day smoked/20) x number of years smoked)).
* Average QTcB or QTcF ≤ 450 msec taken from triplicate assessments at screening; or QTc ≤ 480 msec in subjects with Bundle Branch Block.
* Subject has a post-bronchodilator (400 μg salbutamol) FEV1 of ≥ 35% to ≤ 80% of predicted normal.
* Subject has FEV1/FVC < 0.7 post-bronchodilator (400 μg salbutamol).
* Subjects have a 24hour holter recording that is within normal limits for the individual and does not demonstrate any clinically important abnormality that, in the opinion of the investigator, would make the subject unsuitable for participation in the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject is available to complete all study measurements and procedures.

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the Investigator, may affect subject safety or influence the outcome of the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine and opiates.

The detection of drugs taken for a legitimate medical purpose would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.

* Female subject has a positive pregnancy test.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody (if tested, according to local SOP's).
* History of high alcohol consumption within 1 month of the study defined as:

  * an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof (including allergy to milk protein/lactose) or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Subject has donated a unit (400 mL) of blood within 60 days of screening or, intends to donate during the study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject requires treatment for prostate hypertrophy.
* The subject has a history of narrow angle glaucoma.

Respiratory criteria

* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, pulmonary fibrosis, asthma or any other respiratory condition that might, in the opinion of the Investigator, compromise the safety of the subject or affect the interpretation of the results.
* Subject has poorly controlled COPD, defined as the occurrence of any of the following:

  * Either: acute worsening of COPD that is managed by the subject at home requiring treatment with corticosteroids in the 2 weeks prior to the screening visit.
  * Or: more than two exacerbations in the previous 4 months prior to the screening visit that required a course of oral corticosteroids or, for which the subject was hospitalised.
* Subject has had a respiratory tract infection in the 2 weeks prior to first dose.

Cardiovascular criteria

* Current congestive heart failure (greater than NYHA II) and myocardial infarction (within 9 months of the screening date).
* A history of clinically significant arrhythmia or clinically important 24 h Holter findings that, in the opinion of the Investigator, would cause a safety concern for entry into the study.
* A mean QTc(B) value at screening >450msec, or an ECG that is not suitable for QT measurements (e.g. LBBB or poorly defined termination of the T wave).
* Third degree heart block or pacemaker.
* Risk factors for torsades des pointes (heart failure NYHA II-IV, familial long QT syndrome).
* Elevated resting blood pressure or a mean blood pressure equal to or higher than 150/90 mmHg at screening. A history of and treatment for hypertension is acceptable provided control has been achieved for > 2 months prior to screening.
* A mean heart rate outside the range 50-100 bpm at screening.

Concurrent medication criteria

* Subject requires treatment with nebulised beta-2 agonist or nebulised anticholinergics.
* Subject has received oral or parenteral corticosteroids within 2 weeks of screening.
* Subject is unable to abstain from long-acting bronchodilators from 48 hours prior to the screening and treatment periods (i.e. the last assessment in the dosing period).

(Note, subjects may resume use of their usual medication in between screening and the treatment period if the restrictions in Section 9 Concomitant Medications and Non-Drug Therapies are followed and provided the long acting bronchodilator component is stopped again 48h or more prior to dosing).

* Subject is receiving co-medication with drugs which are commonly recognised to prolong the QTc interval (e.g. quinolones, amiodorane, disopyramide, quinidine, sotalol, chlorpromazine, haloperidol, ketoconazole, terfenadine, cisapride and terodiline).
* Subject requires regular treatment with oral corticosteroids (prednisolone or equivalent).
* Subject is receiving treatment with beta-blockers, except eye drops.
* Subject is receiving treatment with long-term or short-term oxygen therapy, NIPPV or requires nocturnal positive pressure for sleep apnea.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United Kingdom (7):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Waterloo, Liverpool, Merseyside
  - GSK Investigational Site, Clydebank, Glasgow
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Llanishen
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tal-Singer R, Cahn A, Mehta R, Preece A, Crater G, Kelleher D, Pouliquen IJ. Initial assessment of single and repeat doses of inhaled umeclidinium in patients with chronic obstructive pulmonary disease: two randomised studies. Eur J Pharmacol. 2013 Feb 15;701(1-3):40-8. doi: 10.1016/j.ejphar.2012.12.019. Epub 2012 Dec 28. PMID 23276660
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants=par.; umeclidinium=UMEC. A total of 37 unique par. were enrolled in the study; however, 1 par. was randomized and dosed on two separate occasions and is counted as two separate par. on all outputs (thus, 38 par. started study treatment).
Pre-assignment Details: Participants were assigned to one of two cohorts: UMEC 250 micrograms (μg) once daily (QD) or placebo (Cohort 1) and UMEC 1000 μg QD or placebo (Cohort 2) for 7 days. After reporting of Cohorts 1 and 2, it was found that par. in Cohort 2 received UMEC 250 μg in error. Cohort 3 was then recruited, in which par. received UMEC 1000 μg QD or placebo.
Groups:
- Placebo: Participants received either a single inhaled dose or four inhaled doses of matching placebo once daily (QD) for 7 days via a dry powder inhaler (DPI).
- Cohort 1 UMEC 250 µg: Participants received a single inhaled dose of umeclidinium (UMEC) 250 micrograms (µg) formulated with magnesium stearate (MgSt) QD for 7 days via a DPI.
- Cohort 2 UMEC 250 µg in Error: Participants received a single inhaled dose of UMEC 250 μg formulated with MgSt QD for 7 days via a DPI. These participants were to have been randomized to receive UMEC 1000 µg; however, they received UMEC 250 µg in error.
- Cohort 3 UMEC 1000 µg: Participants received four inhaled doses of UMEC 250 μg (equivalent to 1000 μg) formulated with MgSt QD for 7 days via a DPI.
Period: Overall Study
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Started | 9 | 10 (One par. (counted as 2 on outputs) was randomized/dosed with UMEC 250 µg on 2 separate occasions.) | 10 | 9
Completed | 9 | 7 | 9 | 6
Not Completed | 0 | 3 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg | Total
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (4.47) | 63.3 (8.21) | 64.7 (6.31) | 64.2 (7.97) | 64.6 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 4 | 14
  Male | 5 | 6 | 8 | 5 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 9 | 10 | 10 | 9 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any On-treatment Adverse Event (AE) or Any On-treatment Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An on-treatment adverse event is defined as an event that occurred between the start of investigational product and follow-up contact. Refer to the general SAE/non-serious AE module for a complete list of AEs reported in the study. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: From start of treatment to study day 12
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
participants
  Any on-treatment AE | 6 | 2 | 8 | 5
  Any on-treatment SAE | 0 | 0 | 0 | 0

2. Primary Outcome: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) on Days 1 and 7
Description: Blood pressure was measured in a semi-recumbent position at approximately 45 degrees after the participant was kept at rest for at least 5 minutes. SBP and DBP were obtained at pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, and 8 hr post-dose (PD) on Day 1 and at pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, 8 hr, and 24 hr PD on Day 7.
Time Frame: Day 1 (pre-dose and 15 minutes [min], 45 min, 1.5 hours [hr], 4 hr, and 8 hr post-dose) and Day 7 (pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, 8 hr, and 24 hr post-dose)
Population: All Subjects Population (ASP). Only participants with data available at the indicated time points were summarized. Different participants may have been summarized for different parameters/at different time points (reflected by n=X, X, X, X in the category titles), so the overall number of participants summarized reflects everyone in the ASP.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Millimeters of mercury (mmHg)
  SBP, Day 1, pre-dose, n=9, 10, 10, 9 | 138.9 (11.43) | 132.8 (11.97) | 137.4 (10.71) | 138.6 (19.13)
  SBP, Day 1, 15 min PD, n=9, 9, 10, 8 | 135.1 (12.96) | 134.9 (15.05) | 137.7 (9.94) | 135.0 (14.72)
  SBP, Day 1, 45 min PD, n=9, 9, 10, 9 | 133.3 (9.35) | 135.8 (14.63) | 133.9 (11.28) | 140.1 (17.64)
  SBP, Day 1, 1.5 hr PD, n=9, 9, 10, 9 | 140.0 (19.42) | 138.2 (15.79) | 142.1 (12.91) | 145.0 (21.27)
  SBP, Day 1, 4 hr PD, n=9, 9, 10, 9 | 141.0 (15.41) | 139.4 (21.43) | 141.6 (8.86) | 138.9 (11.79)
  SBP, Day 1, 8 hr PD, n=9, 9, 10, 9 | 134.8 (12.22) | 135.7 (15.28) | 140.8 (13.14) | 146.2 (14.19)
  SBP, Day 7, pre-dose, n=9, 7, 9, 6 | 134.3 (9.16) | 131.8 (14.47) | 139.3 (10.59) | 120.2 (10.97)
  SBP, Day 7, 15 min PD, n=9, 7, 9, 6 | 141.3 (13.95) | 134.4 (15.54) | 138.8 (12.67) | 127.5 (14.29)
  SBP, Day 7, 45 min PD, n=9, 7, 9, 6 | 139.7 (13.93) | 135.4 (19.08) | 135.8 (9.28) | 126.3 (14.28)
  SBP, Day 7, 1.5 hr PD, n=9, 7, 9, 6 | 137.8 (15.34) | 141.6 (18.35) | 141.3 (10.9) | 130.2 (10.76)
  SBP, Day 7, 4 hr PD, n=9, 7, 9, 6 | 139.4 (12.91) | 139.6 (15.18) | 141.6 (8.56) | 135.0 (14.6)
  SBP, Day 7, 8 hr PD, n=9, 7, 9, 6 | 136.1 (13.17) | 129.4 (14.32) | 136.1 (13.7) | 125.7 (8.29)
  SBP, Day 7, 24 hr PD, n=9, 7, 9, 6 | 132.1 (9.49) | 135.7 (9.39) | 136.0 (9.82) | 127.5 (7.71)
  DBP, Day 1, pre-dose, n=9, 10, 10, 9 | 81.6 (8.52) | 79.0 (6.69) | 82.1 (7.63) | 82.4 (5.25)
  DBP, Day 1, 15 min PD, n=9, 9, 10, 8 | 79.6 (9.76) | 83.6 (7.47) | 81.4 (7.71) | 85.8 (10.46)
  DBP, Day 1, 45 min PD, n=9, 9, 10, 9 | 78.9 (8.85) | 79.6 (9.58) | 82.8 (9.96) | 83.8 (7.90)
  DBP, Day 1, 1.5 hr PD, n=9, 9, 10, 9 | 79.3 (8.54) | 82.3 (9.26) | 84.0 (6.55) | 85.4 (6.88)
  DBP, Day 1, 4 hr PD, n=9, 9, 10, 9 | 83.4 (11.14) | 81.0 (10.91) | 83.1 (11.13) | 83.7 (6.06)
  DBP, Day 1, 8 hr PD, n=9, 9, 10, 9 | 77.8 (8.67) | 79.9 (8.85) | 80.5 (7.84) | 85.3 (6.08)
  DBP, Day 7, pre-dose, n=9, 7, 9, 6 | 78.7 (8.64) | 82.6 (8.85) | 85.8 (7.79) | 76.5 (4.35)
  DBP, Day 7, 15 min PD, n=9, 7, 9, 6 | 82.8 (11.78) | 82.7 (9.11) | 82.9 (9.29) | 81.8 (5.46)
  DBP, Day 7, 45 min PD, n=9, 7, 9, 6 | 80.6 (10.36) | 81.4 (9.45) | 82.4 (7.04) | 81.8 (6.49)
  DBP, Day 7, 1.5 hr PD, n=9, 7, 9, 6 | 82.2 (9.91) | 82.6 (8.90) | 83.1 (9.97) | 81.7 (3.50)
  DBP, Day 7, 4 hr PD, n=9, 7, 9, 6 | 79.0 (8.97) | 84.0 (7.68) | 83.0 (8.09) | 81.0 (4.00)
  DBP, Day 7, 8 hr PD, n=9, 7, 9, 6 | 76.2 (8.70) | 77.1 (11.51) | 80.7 (7.45) | 77.8 (3.54)
  DBP, Day 7, 24 hr PD, n=9, 7, 9, 6 | 78.2 (8.87) | 81.6 (9.05) | 81.7 (9.70) | 79.8 (4.79)

3. Primary Outcome: Mean Heart Rate (HR) on Days 1 and 7
Description: HR was measured in a semi-recumbent position at approximately 45 degrees after the participant was kept at rest for at least 5 minutes. HR was obtained at pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, and 8 hr post-dose (PD) on Day 1 and at pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, 8 hr, and 24 hr PD on Day 7.
Time Frame: as for outcome 2
Population: All Subjects Population. Only participants with data available at the indicated time points were summarized. Different participants may have been summarized for different parameters/at different time points (reflected by n=X, X, X, X in the category titles), so the overall number of participants summarized reflects everyone in the ASP.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Beats per minute
  Day 1, pre-dose, n=9, 10, 10, 9 | 70.9 (11.09) | 68.3 (10.42) | 72.8 (11.69) | 64.7 (10.34)
  Day 1, 15 min PD, n=9, 9, 10, 8 | 68.2 (10.28) | 67.4 (11.28) | 71.4 (9.86) | 72.3 (13.56)
  Day 1, 45 min PD, n=9, 9, 10, 9 | 66.0 (9.33) | 62.3 (10.90) | 70.2 (11.95) | 66.4 (14.78)
  Day 1, 1.5 hr PD, n=9, 9, 10, 9 | 63.3 (9.42) | 60.7 (12.06) | 65.8 (10.30) | 64.2 (11.05)
  Day 1, 4 hr PD, n=9, 9, 10, 9 | 64.0 (10.37) | 62.0 (10.31) | 70.2 (10.74) | 65.7 (10.20)
  Day 1, 8 hr PD, n=9, 9, 10, 9 | 72.6 (9.93) | 67.4 (9.62) | 77.2 (11.73) | 74.4 (7.35)
  Day 7, pre-dose, n=9, 7, 9, 6 | 70.1 (7.90) | 71.3 (12.64) | 71.4 (14.01) | 69.7 (10.51)
  Day 7, 15 min PD, n=9, 7, 9, 6 | 67.0 (6.61) | 69.4 (12.16) | 68.9 (12.19) | 74.8 (9.39)
  Day 7, 45 min PD, n=9, 6, 9, 6 | 66.8 (9.16) | 66.3 (11.88) | 66.6 (10.98) | 70.0 (10.00)
  Day 7, 1.5 hr PD, n=9, 7, 9, 6 | 65.3 (7.86) | 64.0 (10.92) | 63.8 (8.96) | 67.7 (11.13)
  Day 7, 4 hr PD, n=9, 7, 9, 6 | 64.1 (7.61) | 62.7 (7.74) | 62.6 (9.79) | 67.5 (7.50)
  Day 7, 8 hr PD, n=9, 7, 9, 6 | 74.8 (6.83) | 71.0 (8.60) | 74.8 (8.91) | 73.8 (7.41)
  Day 7, 24 hr PD, n=9, 7, 9, 6 | 73.8 (7.00) | 75.6 (11.50) | 72.6 (8.97) | 70.8 (9.89)

4. Primary Outcome: Maximum and Weighted Mean (0-4 Hour) Heart Rate at Days 1 and 7
Description: Maximum heart rate (Max HR) and weighted mean (WM) from 0-4 hour on Days 1 and 7 were derived. Max HR (0-4 h) is defined as the maximum heart rate attained within 0-4 h. The weighted mean HR (0-4 h) was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. Each of the maximum and weighted mean (0-4h) endpoints for heart rate, was statistically analyzed using a mixed effects model. The terms treatment, baseline, day and any relevant interactions were considered in the model. Least squares means are adjusted for treatment, Baseline, day, treatment by Baseline and Baseline by day interaction, where Baseline is defined as the mean of the three pre-dose assessments.
Time Frame: Day 1 and Day 7
Population: All Subjects Population (ASP). The number of participants presented represent those with data available at the time point being presented; however, all participants in the ASP without missing covariate information are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Beats per minute
  Day 1, Max HR, n=9, 10, 10, 9 | 68.30 (2.009) | 70.56 (1.910) | 71.57 (1.924) | 75.79 (2.066)
  Day 7, Max HR, n=9, 7, 9, 6 | 68.99 (1.917) | 70.24 (2.203) | 66.74 (1.964) | 77.69 (2.398)
  Day 1, WM, n=9, 9, 10, 9 | 63.84 (1.582) | 63.62 (1.584) | 66.17 (1.514) | 70.00 (1.627)
  Day 7, WM, n=9, 7, 9, 6 | 64.83 (1.682) | 64.98 (1.874) | 62.32 (1.698) | 71.89 (2.026)
Statistical Analysis 1: Comparison: Placebo vs Cohort 1 UMEC 250 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [-3.39 to 7.91], Standard Error of Mean 2.777 — Day 1, Max HR
Statistical Analysis 2: Comparison: Placebo vs Cohort 1 UMEC 250 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-4.78 to 7.28], Standard Error of Mean 2.922 — Day 7, Max HR
Statistical Analysis 3: Comparison: Placebo vs Cohort 2 UMEC 250 µg in Error; Test type: Superiority or Other; Mean Difference (Final Values) = 3.27, 95% CI 2-sided [-2.37 to 8.91], Standard Error of Mean 2.772 — Day 1, Max HR
Statistical Analysis 4: Comparison: Placebo vs Cohort 2 UMEC 250 µg in Error; Test type: Superiority or Other; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-7.89 to 3.39], Standard Error of Mean 2.729 — Day 7, Max HR
Statistical Analysis 5: Comparison: Placebo vs Cohort 3 UMEC 1000 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.49, 95% CI 2-sided [1.59 to 13.39], Standard Error of Mean 2.899 — Day 1, Max HR
Statistical Analysis 6: Comparison: Placebo vs Cohort 3 UMEC 1000 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 8.70, 95% CI 2-sided [2.34 to 15.05], Standard Error of Mean 3.079 — Day 7, Max HR
Statistical Analysis 7: Comparison: Placebo vs Cohort 1 UMEC 250 µg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-4.80 to 4.34], Standard Error of Mean 2.243 — Day 1, WM
Statistical Analysis 8: Comparison: Placebo vs Cohort 1 UMEC 250 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-5.09 to 5.40], Standard Error of Mean 2.520 — Day 7, WM
Statistical Analysis 9: Comparison: Placebo vs Cohort 2 UMEC 250 µg in Error; Test type: Superiority or Other; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [-2.12 to 6.77], Standard Error of Mean 2.182 — Day 1, WM
Statistical Analysis 10: Comparison: Placebo vs Cohort 2 UMEC 250 µg in Error; Test type: Superiority or Other; Mean Difference (Final Values) = -2.51, 95% CI 2-sided [-7.48 to 2.45], Standard Error of Mean 2.378 — Day 7, WM
Statistical Analysis 11: Comparison: Placebo vs Cohort 3 UMEC 1000 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.16, 95% CI 2-sided [1.51 to 10.81], Standard Error of Mean 2.282 — Day 1, WM
Statistical Analysis 12: Comparison: Placebo vs Cohort 3 UMEC 1000 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.06, 95% CI 2-sided [1.57 to 12.54], Standard Error of Mean 2.642 — Day 7, WM

5. Primary Outcome: Number of Participants With the Indicated 12-lead Electrocardiogram (ECG) Values on Days 1 and 7
Description: The number of participants with normal (NL), abnormal not clinically significant (Abn NCS), and abnormal clinically significant (Abn CS) ECG findings, as well as those with unavailable results (NA) at pre-dose (PD1, PD2, PD3), and 15 min, 45 min, 1.5 hr, 4 hr, and 8 hr post-dose (PD) on Day 1 and at pre-dose (PD1, PD2, PD3), and 15 min, 45 min, 1.5 hr, 4 hr, 8 hr, and 24 hr post-dose on Day 7 are reported. The following are of potential clinical importance: absolute QTc interval >450 milliseconds (msec); increase from Baseline QTc >60 msec; PR interval <110 and >220 msec; QRS interval <75 and >110 msec. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee.
Time Frame: Day 1 (pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, and 8 hr post-dose) and Day 7 (pre-dose and 15 min, 45 min, 1.5 hr, 4 hr, 8 hr, and 24 hr)
Population: All Subjects Population. Only participants with data available at the indicated time points were summarized.
Measure: Number; unit: Participants
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Participants
  Day 1, PD1, NL, n=9, 10, 10, 9 | 5 | 3 | 6 | 6
  Day 1, PD1, Abn NCS, n=9, 10, 10, 9 | 4 | 7 | 4 | 3
  Day 1, PD1, Abn CS, n=9, 10, 10, 9 | 0 | 0 | 0 | 0
  Day 1, PD1, NA, n=9, 10, 10, 9 | 0 | 0 | 0 | 0
  Day 1, PD2, NL, n=9, 10, 10, 9 | 5 | 3 | 5 | 5
  Day 1, PD2, Abn NCS, n=9, 10, 10, 9 | 4 | 7 | 5 | 3
  Day 1, PD2, Abn CS, n=9, 10, 10, 9 | 0 | 0 | 0 | 0
  Day 1, PD2, NA, n=9, 10, 10, 9 | 0 | 0 | 0 | 1
  Day 1, PD3, NL, n=9, 10, 10, 9 | 4 | 4 | 5 | 5
  Day 1, PD3, Abn NCS, n=9, 10, 10, 9 | 5 | 6 | 5 | 3
  Day 1, PD3, Abn CS, 9, 10, 10, 9 | 0 | 0 | 0 | 0
  Day 1, PD3, NA, n=9, 10, 10, 9 | 0 | 0 | 0 | 1
  Day 1, 15 min PD, NL, n=9, 9, 10, 9 | 4 | 3 | 7 | 6
  Day 1, 15 min PD, Abn NCS, n=9, 9, 10, 9 | 5 | 6 | 3 | 3
  Day 1, 15 min PD, Abn CS, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 15 min PD, NA, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 45 min PD, NL, n=9, 9, 10, 9 | 5 | 3 | 7 | 6
  Day 1, 45 min PD, Abn NCS, n=9, 9, 10, 9 | 4 | 6 | 3 | 3
  Day 1, 45 min PD, Abn CS, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 45 min PD, NA, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 1.5 hr PD, NL, n=9, 9, 10, 9 | 5 | 6 | 6 | 5
  Day 1, 1.5 hr PD, Abn NCS, n=9, 9, 10, 9 | 4 | 3 | 4 | 4
  Day 1, 1.5 hr PD, Abn CS, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 1.5 hr PD, NA, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 4 hr PD, NL, n=9, 9, 10, 9 | 4 | 4 | 6 | 5
  Day 1, 4 hr PD, Abn NCS, n=9, 9, 10, 9 | 5 | 5 | 4 | 4
  Day 1, 4 hr PD, Abn CS, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 4 hr PD, NA, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 8 hr PD, NL, n=9, 9, 10, 9 | 5 | 6 | 7 | 6
  Day 1, 8 hr PD, Abn NCS, n=9, 9, 10, 9 | 4 | 3 | 3 | 3
  Day 1, 8 hr PD, Abn CS, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 1, 8 hr PD, NA, n=9, 9, 10, 9 | 0 | 0 | 0 | 0
  Day 7, PD1, NL, n=9, 7, 9, 6 | 4 | 4 | 7 | 3
  Day 7, PD1, Abn NCS, n=9, 7, 9, 6 | 5 | 3 | 2 | 3
  Day 7, PD1, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, PD1, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, PD2, NL, n=9, 7, 8, 6 | 4 | 4 | 6 | 3
  Day 7, PD2, Abn NCS, n=9, 7, 8, 6 | 5 | 3 | 2 | 3
  Day 7, PD2, Abn CS, n=9, 7, 8, 6 | 0 | 0 | 0 | 0
  Day 7, PD2, NA, n=9, 7, 8, 6 | 0 | 0 | 0 | 0
  Day 7, PD3, NL, n=9, 7, 8, 6 | 4 | 3 | 6 | 3
  Day 7, PD3, Abn NCS, n=9, 7, 8, 6 | 5 | 4 | 2 | 3
  Day 7, PD3, Abn CS, 9, 7, 8, 6 | 0 | 0 | 0 | 0
  Day 7, PD3, NA, n=9, 7, 8, 6 | 0 | 0 | 0 | 0
  Day 7, 15 min PD, NL, n=9, 7, 9, 6 | 4 | 4 | 7 | 3
  Day 7, 15 min PD, Abn NCS, n=9, 7, 9, 6 | 5 | 3 | 2 | 3
  Day 7, 15 min PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 15 min PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 45 min PD, NL, n=9, 7, 9, 6 | 4 | 4 | 6 | 3
  Day 7, 45 min PD, Abn NCS, n=9, 7, 9, 6 | 5 | 3 | 3 | 3
  Day 7, 45 min PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 45 min PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 1.5 hr PD, NL, n=9, 7, 9, 6 | 4 | 4 | 7 | 3
  Day 7, 1.5 hr PD, Abn NCS, n=9, 7, 9, 6 | 5 | 3 | 2 | 3
  Day 7, 1.5 hr PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 1.5 hr PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 4 hr PD, NL, n=9, 7, 9, 6 | 5 | 5 | 7 | 3
  Day 7, 4 hr PD, Abn NCS, n=9, 7, 9, 6 | 4 | 2 | 2 | 3
  Day 7, 4 hr PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 4 hr PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 8 hr PD, NL, n=9, 7, 9, 6 | 4 | 4 | 7 | 3
  Day 7, 8 hr PD, Abn NCS, n=9, 7, 9, 6 | 5 | 3 | 2 | 3
  Day 7, 8 hr PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 8 hr PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 24 hr PD, NL, n=9, 7, 9, 6 | 4 | 2 | 6 | 3
  Day 7, 24 hr PD, Abn NCS, n=9, 7, 9, 6 | 5 | 5 | 3 | 3
  Day 7, 24 hr PD, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 0 | 0
  Day 7, 24 hr PD, NA, n=9, 7, 9, 6 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal 24-hour Holter Findings at Screening and Day 7
Description: Twenty-four hour Holter ECG values were obtained at Screening and on Day 7. During the Screening procedure and study, standard Holter monitors were used (in order to exclude participants with underlying cardiac arrhythmogenicity). During the treatment periods, Holter monitors were only switched on immediately prior to dosing (up to 15 minutes pre-dose) so as to capture Holter ECG data from the 24 hour period following dosing. The following summary data were transcribed into the Case Report Form: Maximum and mean (0 to24 hour) heart rate; normal and aberrant beats and arrhythmias. Analysis of the Holter tapes was arranged by GlaxoSmithKline.The number of participants with normal (NL), abnormal not clinically significant (Abn NCS), and abnormal clinically significant (Abn CS) ECG findings, as well as those with unavailable results (NA) at Screening and Day 7, are reported. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee.
Time Frame: Screening and Day 7
Population: All Subjects Population. Only participants with data available at the indicated time points were summarized.
Measure: Number; unit: Participants
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Participants
  Screening, NL, n=9 ,10, 10, 9 | 2 | 6 | 5 | 3
  Screening, Abn NCS, n=9 ,10, 10, 9 | 7 | 4 | 4 | 5
  Screening, Abn CS, n=9 ,10, 10, 9 | 0 | 0 | 1 | 1
  Day7, NL, n=9, 7, 9, 6 | 3 | 3 | 2 | 1
  Day7, Abn NCS, n=9, 7, 9, 6 | 6 | 3 | 6 | 5
  Day7, Abn CS, n=9, 7, 9, 6 | 0 | 0 | 1 | 0
  Day7, NA, n=9, 7, 9, 6 | 0 | 1 | 0 | 0

7. Primary Outcome: Maximum and Mean (0-24 Hour) Heart Rate From Holter Monitoring on Day 7
Description: Maximum heart rate (Max HR) and mean HR from 0-24 hour Holter monitoring on treatment Day 7 were derived. The analysis was adjusted for treatment and Baseline, where Baseline is defined as the corresponding summary measure (i.e., mean heart rate [0-24 hours] or maximum heart rate [0-24 hours]) from screening records.
Time Frame: Day 7
Population: All Subjects Population. The number of participants presented represent those with data available at the time point being presented; however, all participants in the ASP without missing covariate information are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 6 | 9 | 6
Beats per minute
  Max HR | 125.19 (4.744) | 134.08 (5.810) | 127.48 (4.724) | 126.91 (5.785)
  Mean HR | 77.47 (1.896) | 75.94 (2.306) | 75.96 (1.888) | 76.75 (2.312)

8. Primary Outcome: Mean Forced Expiratory Volume in One Second (FEV1) at Screening and on Days 1 and 7
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured at Screening, pre-dose, and 4 hours (hr) post-dose on Day 1 and Day 7. FEV1 tests were repeated until three technically acceptable measurements were made.
Time Frame: Screening, Day 1, and Day 7
Population: All Subjects Population. Only participants with data available at the indicated time points were summarized.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Liters
  Screening, n=9, 10, 10, 9 | 1.556 (0.6315) | 1.253 (0.4338) | 1.562 (0.5066) | 1.364 (0.3504)
  Day 1, pre-dose, n=9, 10, 10, 9 | 1.294 (0.4642) | 1.059 (0.3509) | 1.443 (0.4840) | 1.289 (0.2968)
  Day 1, 4 hr post-dose, n=9, 9, 10, 9 | 1.309 (0.4333) | 1.250 (0.3934) | 1.565 (0.5858) | 1.534 (0.3389)
  Day 7, pre-dose, n=9, 7, 9, 6 | 1.263 (0.4695) | 1.153 (0.4066) | 1.593 (0.5425) | 1.483 (0.3055)
  Day 7, 4 hr post-dose, n=9, 7, 9, 6 | 1.250 (0.5143) | 1.181 (0.3875) | 1.564 (0.5476) | 1.517 (0.2685)

9. Primary Outcome: Total Number of Salbutamol Doses Taken Over the 7 -Day Study Period
Description: The total number of salbutamol doses taken per day was recorded by the participants in their dairy card over the entire 7-day treatment period. Diaries were reviewed by the Investigator when participants were admitted to the unit on Day 1, Day 7, and Day 8. Salbutamol was given as rescue medication, defined as a quick-relief or fast-acting medication that is given in addition to the investigational drug or placebo that can alleviate symptoms due to disease or lack of efficacy of the study treatment.
Time Frame: Day 1 to Day 7
Population: All Subjects Population. Only those participants who took at least one dose of salbutamol were summarized.
Measure: Number; unit: salbutamol doses
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 6 | 3 | 5 | 5
salbutamol doses | 18 | 33 | 33 | 29

10. Primary Outcome: Albumin, Total Protein, Hemoglobin, and Mean Corpuscle Hemoglobin Concentration (MCHC) Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of albumin, total protein, hemoglobin, and MCHC values pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Grams per liter (G/L)
  Albumin, Day 1, n=9, 9, 10, 9 | 42.3 (3.43) | 43.9 (2.09) | 43.7 (2.16) | 44.1 (3.10)
  Albumin, Day 7, n=8, 7, 9, 6 | 43.1 (1.81) | 44.0 (1.15) | 43.8 (2.64) | 44.0 (2.61)
  Total protein, Day 1, n=9, 9, 10, 9 | 69.4 (5.48) | 70.0 (3.24) | 69.9 (3.70) | 69.8 (3.46)
  Total protein, Day 7, n=8, 7, 9, 6 | 68.6 (3.16) | 70.0 (2.16) | 71.0 (4.53) | 69.7 (3.83)
  Hemoglobin, Day 1, n=9, 9, 10, 9 | 152.2 (8.60) | 148.0 (14.19) | 147.4 (11.84) | 145.4 (16.18)
  Hemoglobin, Day 7, n=9, 6, 9, 6 | 151.4 (7.80) | 145.8 (14.77) | 147.4 (13.71) | 143.5 (16.61)
  MCHC, Day 1, n=9, 9, 10, 9 | 340.0 (6.10) | 338.7 (5.39) | 339.9 (5.49) | 337.2 (3.63)
  MCHC, Day 7, n=9, 6, 9, 6 | 337.6 (7.84) | 340.7 (5.20) | 337.4 (5.59) | 337.3 (5.20)

11. Primary Outcome: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT) Values on Day1 and Day 7
Description: Blood samples were collected for the measurement of ALP, ALT, AST, and GGT Pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
International units per liter (IU/L)
  ALP, Day 1, n=9, 9, 10, 9 | 74.0 (20.20) | 76.8 (15.11) | 69.0 (18.43) | 63.8 (20.00)
  ALP, Day 7, n=8, 7, 9, 6 | 71.6 (20.18) | 73.1 (16.16) | 71.1 (16.47) | 67.7 (18.15)
  ALT, Day 1, n=9, 9, 10, 9 | 15.6 (10.36) | 15.6 (6.06) | 24.2 (9.66) | 18.6 (9.49)
  ALT, Day 7, n=8, 7, 9, 6 | 15.9 (6.85) | 15.6 (7.11) | 29.8 (12.81) | 20.7 (9.85)
  AST, Day 1, n=9, 9, 10, 9 | 20.9 (5.90) | 18.9 (3.48) | 26.5 (10.28) | 22.6 (8.65)
  AST, Day 7, n=8, 7, 9, 6 | 19.3 (6.16) | 19.4 (4.31) | 30.7 (12.16) | 25.2 (8.18)
  GGT, Day 1, n=9, 9, 10, 9 | 31.3 (20.62) | 28.0 (13.19) | 61.0 (56.20) | 37.7 (31.25)
  GGT, Day 7, n=8, 7, 9, 6 | 29.9 (18.88) | 24.7 (6.78) | 66.0 (68.81) | 39.8 (32.73)

12. Primary Outcome: Direct Bilirubin, Total Bilirubin, and Creatinine Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of direct bilirubin, total bilirubin, and creatinine at pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Groups:
- Cohort 2 UMEC 250 µg in Error: Participants received a single inhaled dose of UMEC19 250 μg formulated with MgSt QD for 7 days via a DPI. These participants were to have been randomized to receive UMEC 1000 µg; however, they received UMEC 250 µg in error.
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Micromoles per liter (µmol/L)
  Direct bilirubin, Day 1, n=6, 9, 10 | 2.3 (1.97) | 1.7 (0.50) | 2.0 (1.15) | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, Cohort 3 data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Direct bilirubin, Day 7, n=5, 7, 9 | 2.0 (1.41) | 2.0 (0.58) | 2.2 (0.67) | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, Cohort 3 data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Total bilirubin, Day 1, n=9, 9, 10, 9 | 10.8 (4.44) | 8.2 (1.20) | 10.9 (4.01) | 10.2 (3.03)
  Total bilirubin, Day 7, n=8, 7, 9, 6 | 9.3 (4.03) | 9.9 (2.27) | 10.8 (3.11) | 11.0 (3.16)
  Creatinine, Day 1, n=9, 9, 10, 9 | 76.2 (12.15) | 84.3 (15.64) | 80.1 (14.26) | 87.0 (33.59)
  Creatinine, Day 7, n=8, 7, 9, 6 | 78.8 (10.53) | 80.1 (14.37) | 82.6 (12.83) | 93.0 (39.80)

13. Primary Outcome: Calcium, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of calcium, glucose, potassium, sodium, and urea/BUN pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
Millimoles per liter (mmol/L)
  Calcium, Day 1, n=9, 9, 10, 9 | 2.317 (0.0622) | 2.329 (0.0697) | 2.342 (0.1215) | 2.311 (0.0807)
  Calcium, Day 7, n=8, 7, 9, 6 | 2.320 (0.0454) | 2.321 (0.0308) | 2.370 (0.1411) | 2.343 (0.0631)
  Glucose, Day 1, n=9, 9, 10, 9 | 5.16 (0.937) | 5.13 (0.524) | 5.38 (0.751) | 5.26 (0.921)
  Glucose, Day 7, n=8, 7, 9, 6 | 5.25 (0.746) | 5.10 (0.792) | 5.84 (0.948) | 5.42 (0.717)
  Potassium, Day 1, n=9, 9, 10, 9 | 4.67 (0.472) | 4.70 (0.485) | 4.50 (0.579) | 4.36 (0.364)
  Potassium, Day 7, n=8, 7, 9, 6 | 4.58 (0.276) | 4.74 (0.431) | 4.48 (0.519) | 4.45 (0.428)
  Sodium, Day 1, n=9, 9, 10, 9 | 138.8 (2.59) | 140.6 (1.51) | 140.6 (2.27) | 139.6 (1.59)
  Sodium, Day 7, n=8, 7, 9, 6 | 140.4 (2.88) | 140.0 (1.15) | 140.2 (2.44) | 139.2 (2.40)
  Urea/BUN, Day 1, n=9, 9, 10, 9 | 4.92 (1.730) | 5.29 (0.842) | 5.77 (1.854) | 5.72 (2.440)
  Urea/BUN, Day 7, n=8, 7, 9, 6 | 5.15 (1.032) | 5.51 (0.691) | 5.70 (1.562) | 5.88 (3.020)

14. Primary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, Total Neutrophil (ANC: Absolute Neutrophil Count), Platelet, and White Blood Cell (WBC) Count Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils (ANC), platelets, and white blood cell (WBC) count pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
10^9 cells per liter (GI/L)
  Basophils, Day 1, n=9, 9, 10, 9 | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Basophils, Day 7, n=9, 6, 9, 6 | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Eosinophils, Day 1, n=9, 9, 10, 9 | 0.248 (0.1052) | 0.319 (0.1968) | 0.352 (0.2951) | 0.144 (0.0910)
  Eosinophils, Day 7, n=9, 6, 9, 6 | 0.232 (0.0793) | 0.280 (0.1754) | 0.312 (0.2672) | 0.153 (0.0911)
  Lymphocytes, Day 1, n=9, 9, 10, 9 | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Lymphocytes, Day 7, n=9, 6, 9, 6 | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed. | NA (NA) — Per protocol, data were collected for participants in all 3 cohorts; however, data were not fully reported to GSK by the vendor. This oversight was recently detected, and this summary will be amended once remedial work has been completed.
  Monocytes, Day 1, n=9, 9, 10, 9 | 0.510 (0.1348) | 0.614 (0.3648) | 0.607 (0.1594) | 0.506 (0.2010)
  Monocytes, Day 7, n=9, 6, 9, 6 | 0.448 (0.1313) | 0.562 (0.2791) | 0.657 (0.1993) | 0.503 (0.2430)
  ANC, Day 1, n=9, 9, 10, 9 | 5.233 (2.0968) | 5.306 (1.3061) | 4.244 (1.3332) | 4.946 (2.3879)
  ANC, Day 7, n=9, 6, 9, 6 | 4.706 (1.8634) | 5.023 (1.4969) | 4.067 (1.0184) | 5.323 (1.8539)
  Platelets, Day 1, n=9, 9, 10, 9 | 278.1 (66.25) | 238.2 (39.71) | 254.7 (51.04) | 222.4 (43.16)
  Platelets, Day 7, n=9, 6, 9, 6 | 271.8 (53.73) | 256.8 (36.71) | 255.1 (61.42) | 250.3 (59.37)
  WBC count, Day 1, n=9, 9, 10, 9 | 8.06 (2.220) | 8.52 (2.153) | 7.11 (1.692) | 7.56 (2.572)
  WBC count, Day 7, n=9, 6, 9, 6 | 7.49 (2.211) | 8.15 (2.519) | 7.13 (1.564) | 7.87 (2.067)

15. Primary Outcome: Mean Corpuscle Hemoglobin (MCH) Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of MCH pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: picograms/cell (pg)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
picograms/cell (pg)
  Day 1, n=9, 9, 10, 9 | 31.92 (1.711) | 32.44 (2.371) | 31.25 (1.978) | 31.70 (1.859)
  Day 7, n=9, 6, 9, 6 | 31.71 (1.661) | 32.20 (2.871) | 31.22 (1.999) | 31.95 (2.146)

16. Primary Outcome: Mean Corpuscle Volume (MCV) Values on Day 1 and Day 7
Description: Blood samples were collected for the measurement of MCV pre-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^-15 liters (femtoliters)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 9 | 10 | 10 | 9
10^-15 liters (femtoliters)
  Day 1, n=9, 9, 10, 9 | 93.9 (3.66) | 95.9 (7.06) | 91.9 (4.93) | 94.0 (5.32)
  Day 7, n=9, 6, 9, 6 | 94.0 (3.50) | 94.5 (7.12) | 92.6 (5.34) | 94.8 (5.49)

17. Secondary Outcome: Mean AUC(0-2), AUC(0-8), and AUC(0-t) of UMEC on Day 1 and Day 7
Description: Area under the concentration-time (AUC) curve from time zero (pre-dose) to 2 hours (AUC[0-2]), from time zero to 8 hours (AUC[0-8]), from time zero to the last time of a quantifiable concentration of UMEC (AUC[0-t]) on Day 1 and Day 7 were measured. AUC is a measure of systemic exposure. Blood samples were collected pre-dose and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose on Day 1 and Day 7. Also, a 24 hr blood sample was collected on Day 7.
Time Frame: Day 1 and Day 7: pre-dose, and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose; 24 hr post-dose on Day 7
Population: Pharmacokinetic (PK) Population: participants (par.) in the ASP for whom a PK sample was obtained and analyzed. Different par. may have been summarized for different parameters/at different time points (reflected by n=X, X, X, X in the category titles), so the overall number of par. summarized reflects everyone in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr * nanograms per milliliter (ng/mL)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
hr * nanograms per milliliter (ng/mL)
  AUC(0-2), Day 1, n=0, 8, 9, 9 |  | 0.19675 (19.7) | 0.08134 (108.0) | 0.95719 (233.2)
  AUC(0-2), Day 7, n=0, 6, 8, 6 |  | 0.31951 (51.6) | 0.15527 (66.5) | 1.92508 (31.1)
  AUC(0-8), Day 1, n=0, 0, 0, 9 |  | NA (NA) — Due to non-quantifiable data at the lower dose (250 µg) at later time points, data for this parameter could not be calculated. | NA (NA) — Due to non-quantifiable data at the lower dose (250 µg) at later time points, data for this parameter could not be calculated. | 2.029 (69.8)
  AUC(0-8), Day 7, n=0, 0, 0, 6 |  | NA (NA) — Due to non-quantifiable data at the lower dose (250 µg) at later time points, data for this parameter could not be calculated. | NA (NA) — Due to non-quantifiable data at the lower dose (250 µg) at later time points, data for this parameter could not be calculated. | 3.320 (33.3)
  AUC(0-t), Day 1, n=0, 8, 9, 9 |  | 0.26071 (39.1) | 0.03614 (1707.8) | 0.93299 (5820.5)
  AUC(0-t), Day 7, n=0, 6, 8, 6 |  | 0.55514 (113.2) | 0.30526 (134.3) | 4.86204 (42.8)

18. Secondary Outcome: Cmax of UMEC on Day 1 and Day 7
Description: Cmax is defined as the maximum observed concentration of UMEC and was measured on Day 1 and Day 7. Blood samples were collected pre-dose and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose on Day 1 and Day 7. Also, a 24 hr blood sample was collected on Day 7.
Time Frame: Day 1 and Day 7: pre-dose, and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose; 24 hr post-dose on Day 7
Population: PK Population. Only participants with data available at the indicated time points were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
nanograms per milliliter (ng/mL)
  Day 1, n=0, 8, 9, 9 |  | 0.21654 (32.0) | 0.07915 (147.6) | 1.52835 (53.6)
  Day 7, n=0, 6, 8, 6 |  | 0.33206 (58.3) | 0.16448 (74.2) | 2.75864 (60.5)

19. Secondary Outcome: Tmax and Tlastof UMEC on Day 1 and Day 7
Description: Tmax is defined as the time to reach the observed maximum concentration, and tlast is defined as the time of the last quantifiable concentration of UMEC; both were measured on Day 1 and Day 7. Blood samples were collected pre-dose, and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose on Day 1 and Day 7. Also, a 24 hr blood sample was collected on Day 7.
Time Frame: Day 1 and Day 7: pre-dose, and 5 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose; 24 hr post-dose on Day 7
Population: PK Population. Only participants with data available at the indicated time points were summarized. Different participants may have been summarized for different parameters/at different time points (reflected by n=X, X, X, X in the category titles), so the overall number of participants summarized reflects everyone in the PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
hours
  tmax, Day 1, n=0, 8, 8, 9 |  | 0.080 [0.08 to 0.50] | 0.250 [0.08 to 0.28] | 0.250 [0.08 to 0.28]
  tmax, Day 7, n=0, 6, 8, 6 |  | 0.080 [0.02 to 0.25] | 0.165 [0.08 to 0.32] | 0.240 [0.07 to 0.25]
  tlast, Day 1, n=0, 8, 8, 9 |  | 4.000 [2.00 to 8.12] | 2.000 [0.08 to 4.00] | 8.000 [0.08 to 8.00]
  tlast, Day 7, n=0, 6, 8, 6 |  | 6.000 [2.00 to 27.05] | 6.015 [2.00 to 24.00] | 24.010 [24.00 to 24.48]

20. Secondary Outcome: Ae(0-4), Ae(0-8), Ae(0-12), and Ae(0-24) of UMEC on Day 1 and Day 7
Description: Urinary recovery of unchanged drug (UMEC) within the first 8, 12, and 24 hours (Ae[0-8], Ae[0-12], and Ae[0-24], respectively) on Day 1 and within the first 4, 8, 12, and 24 hours (Ae[0-4], Ae[0-8], Ae[0-12], and Ae[0-24], respectively) on Day 7 was estimated. Urine samples were collected from 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1 and from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7.
Time Frame: From 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1; from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
nanograms (ng)
  Ae(0-4), Day 7, n=0, 5, 8, 6 |  | 1223.6 (77.8) | 669.5 (129.8) | 11854.5 (65.8)
  Ae(0-8), Day 1, n=0, 6, 7, 8 |  | 1756.0 (46.6) | 755.9 (101.5) | 13435.9 (53.8)
  Ae(0-8), Day 7, n=0, 5, 8, 6 |  | 3115.8 (27.2) | 1430.8 (49.6) | 19319.3 (50.5)
  Ae(0-12), Day 1, n=0, 6, 7, 8 |  | 2022.3 (41.2) | 921.7 (97.6) | 16069.2 (56.0)
  Ae(0-12), Day 7, n=0, 5, 8, 6 |  | 4165.6 (15.3) | 1960.5 (53.6) | 23496.1 (44.7)
  Ae(0-24), Day 1, n=0, 6, 7, 8 |  | 2503.5 (38.0) | 1420.3 (130.9) | 19552.7 (47.4)
  Ae(0-24), Day 7, n=0, 5, 8, 6 |  | 5606.2 (15.3) | 2984.5 (52.9) | 32140.0 (36.2)

21. Secondary Outcome: Fe(0-4), Fe(0-8), Fe(0-12), and Fe(0-24) of UMEC on Day 1 and Day 7
Description: The fraction of the total dose excreted (Fe) in each interval was estimated as the urinary recovery of unchanged drug (Ae) per dose. Urine samples were collected from 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1 and from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7.
Time Frame: From 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1; from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7
Population: PK Population: Only participants with data available at the indicated time points were summarized. Different participants may have been summarized for different parameters/at different time points (reflected by n=X, X, X, X in the category titles), so the overall number of participants summarized reflects everyone in the PK Population.
Measure: Mean (Standard Deviation); unit: Percentage of dose administered
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
Percentage of dose administered
  Fe(0-4), Day 7, n=0, 5, 8, 6 |  | 0.58 (0.35) | 0.37 (0.30) | 1.35 (0.70)
  Fe(0-8), Day 1, n=0, 6, 8, 8 |  | 0.76 (0.35) | 0.34 (0.28) | 1.49 (0.68)
  Fe(0-8), Day 7, n=0, 5, 8, 6 |  | 1.28 (0.30) | 0.62 (0.26) | 2.10 (0.84)
  Fe(0-12), Day 1, n=0, 6, 8, 8 |  | 0.87 (0.38) | 0.41 (0.32) | 1.78 (0.77)
  Fe(0-12), Day 7, n=0, 5, 8, 6 |  | 1.68 (0.25) | 0.86 (0.36) | 2.52 (0.99)
  Fe(0-24), Day 1, n=0, 6, 8, 8 |  | 1.06 (0.41) | 0.70 (0.61) | 2.12 (0.82)
  Fe(0-24), Day 7, n=0, 5, 8, 6 |  | 2.26 (0.33) | 1.31 (0.54) | 3.38 (1.15)

22. Secondary Outcome: Renal Clearance of UMEC on Day 1 and Day 7
Description: Renal clearance was calculated as the urinary recovery of unchanged drug from time zero to time x (Ae[0-x])/area under concentration from time zero to time x (AUC[0-x]) for the longest period of time after dosing when both could be accurately determined (where x is either 8, 12, or 24). Urine samples were collected from 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1 and from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7.
Time Frame: From 0-8 hours (hr), 8-12 hr, and 12-24 hr on Day 1; from 0-4 hr, 4-8 hr, 8-12 hr, and 12-24 hr on Day 7
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/hr)
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 8 | 9 | 9
Liters/hour (L/hr)
  Day 1, n=0, 1, 0, 8 |  | 6.5229 (NA) — A dispersion cannot be calculated for a single participant. | NA (NA) — Due to non-quantifiable data at the lower dose (250 µg) at later time points, data for this parameter could not be calculated. | 5.6173 (39.5)
  Day 7, n=0, 4, 6, 6 |  | 2.5923 (103.6) | 4.0826 (19.3) | 6.6104 (33.1)

23. Secondary Outcome: Urine Half Life (t1/2) of UMEC on Day 7
Description: Urine half life (t1/2) of UMEC on Day 7 was estimated. Urine samples were collected from 0-4 hours (hr), 4-8 hr, 8-12 hr, and 12-24 hr on Day 7.
Time Frame: From 0-4 hours (hr), 4-8 hr, 8-12 hr, and 12-24 hr on Day 7
Population: PK Population. Only participants with data available at the indicated time points were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Number analyzed (Participants) | 0 | 2 | 4 | 4
hours |  | 5.785 (39.4) | 8.299 (37.3) | 7.643 (33.4)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs (events occurring between the start of investigational product and follow-up contact) were collected from the start of study medication to the end of the treatment period (up to study day 12).
Description: On-treatment SAEs and non-serious AEs were collected in members of the All Subjects Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | Cohort 1 UMEC 250 µg | Cohort 2 UMEC 250 µg in Error | Cohort 3 UMEC 1000 µg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 6/9 | 2/10 | 8/10 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Cohort 1 UMEC 250 µg (N=10) | Cohort 2 UMEC 250 µg in Error (N=10) | Cohort 3 UMEC 1000 µg (N=9)
Headache (Nervous system disorders) | 1 | 1 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Absess jaw (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Subject 303 and Subject 317 correspond to the same participant who was randomized and dosed on two separate occasions. This participant has been counted as two separate participants on all the outputs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.